CLINICAL TRIAL: NCT00150891
Title: Role of Th1, Th2 and Monokine Responses as Risk Factors of Acute and Chronic Renal Transplant Rejection - Impact of Different Immunosuppressive Protocols
Brief Title: Th1, Th2 and Monokine Responses as Risk Factors of Renal Transplant Rejection
Status: Completed | Type: Observational
Sponsor: University of Giessen (Other)
Collaborators: Heidelberg University (Other); Astellas Pharma Inc (Industry); Novartis (Industry); Fresenius AG (Industry); Hoffmann-La Roche (Industry); Biotest (Industry)
Other Study IDs: NTx-prosp-001
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2007-05-10 (Estimated); Status verified 2007-05

CONDITIONS: Renal Failure, Chronic
Keywords: Th1; Th2; B cell; monokines; kidney transplantation; acute rejection; chronic rejection
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Kidney Transplantation; Cyclosporine; Tacrolimus; Azathioprine; Mycophenolic Acid

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Kidney transplantation
Drug: cyclosporine A
Drug: tacrolimus
Drug: azathioprine
Drug: mycophenolate mofetil

SUMMARY:
Chronic transplant rejection remains the main cause of late kidney graft loss. We showed previously that patients with pretransplant CD4 helper defects and low in-vitro IL-10 responses demonstrated an extremely low risk of acute rejection and a significantly better 1- and 3-year graft function whereas pretransplant Th1 responses were not predictive (Weimer R et al. 1996 and 1998). In liver transplant recipients, we found CD4 helper function and in-vitro IL-10 responses significantly decreased compared to CsA-treated patients (Zipperle et al. 1997). If the same effect will be demonstrated in renal transplant recipients, Tacrolimus (Tacr) treatment might result in enhanced graft survival compared to CsA, when CD4 helper function and in-vitro IL-10 responses of the individual patient are elevated. Other studies of our group suggest a beneficial role of enhanced T-suppressor activity and of an IL-6 independent B cell/monocyte defect in the maintenance of long-term stable graft function, whereas enhanced monokine secretion (TNF-a, GM-CSF, IL-6) was found in chronic rejection (Weimer et al. 1990, 1992, 1994, 1998).

In the current randomized prospective study we will analyze the impact of CsA versus Tacr and of MMF versus azathioprine on Th1, Th2 and monokine responses and their predictive value regarding occurrence of acute and chronic rejection. With a proposed follow-up of 5 years this study might enable a patient-tailored immunosuppressive therapy resulting in prolonged graft survival.

DETAILED DESCRIPTION:
Chronic transplant rejection remains the main cause of late kidney graft loss. We showed previously that patients with pretransplant CD4 helper defects and low in-vitro IL-10 responses demonstrated an extremely low risk of acute rejection and a significantly better 1- and 3-year graft function whereas pretransplant Th1 responses were not predictive (Weimer R et al. 1996 and 1998). In liver transplant recipients, we found CD4 helper function and in-vitro IL-10 responses significantly decreased compared to CsA-treated patients (Zipperle et al. 1997). If the same effect will be demonstrated in renal transplant recipients, Tacrolimus (Tacr) treatment might result in enhanced graft survival compared to CsA, when CD4 helper function and in-vitro IL-10 responses of the individual patient are elevated. Other studies of our group suggest a beneficial role of enhanced T-suppressor activity and of an IL-6 independent B cell/monocyte defect in the maintenance of long-term stable graft function, whereas enhanced monokine secretion (TNF-a, GM-CSF, IL-6) was found in chronic rejection (Weimer et al. 1990, 1992, 1994, 1998).

In the current randomized prospective study we will analyze the impact of CsA versus Tacr and of MMF versus azathioprine (Aza; 3 treatment groups: CsA/Aza, CsA/MMF and Tacr/Aza; steroid and prophylactic ATG treatment according to the Giessen protocol) on immune parameters and their predictive value regarding occurrence of acute and chronic rejection. As immune parameters we will assess CD4 helper function, in-vitro IL-4 and IL-10 responses of T cells and CD4+ T cells, respectively, in allogeneic cocultures of patient T cells with control B cells and in PHA-stimulated T cell cultures, T-cell dependent (PWM-stimulated allogeneic cocultures) and T-independent (SAC I-stimulated B cell cultures) immunoglobulin-secreting cell (ISC) responses, B-cell IL-6 and IL-10 responses and monokine responses (LPS-stimulated monocyte cultures) pretransplant, and 4 months, 1 year, 2 years and 5 years posttransplant. Serum cytokines and easily measurable parameters as neopterin, sIL-1RA and sCD30 will be assessed at the same time points. The same is true for flow cytometric analysis of cytokine receptor, adhesion molecule, costimulator molecule and surface molecule expression, respectively, which play an important role in cell-cell interactions and tolerance induction. Cytokine promoter gene polymorphisms will be determined to potentially enable pretransplant risk estimation. To establish a broadly available and rapid diagnostic method, we will compare the data of intracellular cytokine testing with the results of the much more difficult and time consuming coculture analyses used in our previous studies.

With a proposed follow-up of 5 years this prospective randomized study might enable a patient-tailored immunosuppressive therapy resulting in better graft function and prolonged graft survival by preventing chronic allograft rejection.

Weimer R, Pomer S, Staehler G, Opelz G. Increased T suppressor activity in renal transplant recipients with long-term stable graft function. Clinical Transplantation 1990; 4: 280-286

Weimer R, Zipperle S, Daniel V, Pomer S, Staehler G, Opelz G. In vitro B cell response in long-term renal transplant recipients. Transplant Proc 1992; 24(6): 2537-2538

Weimer R, Zipperle S, Daniel V, Pomer S, Staehler G, Opelz G. IL-6 independent monocyte/B cell defect in renal transplant recipients with long-term stable graft function. Transplantation 1994; 57(1): 54-59

Weimer R, Zipperle S, Daniel V, Carl S, Staehler G, Opelz G. Pretransplant CD4 helper function and IL-10 response predict risk of acute kidney graft rejection. Transplantation 1996; 62(11): 1606-1614

Zipperle S, Weimer R, Golling M, Daniel V, Otto G, Opelz G. Impaired T cell IL-10 secretion and CD4 helper function in liver transplant patients treated with tacrolimus. Transplant Proc 1997; 29(1-2): 1079-1080

Weimer R, Zipperle S, Daniel V, Carl S, Staehler G, Opelz G. Superior 3-year kidney graft function in patients with impaired pretransplant Th2 responses. Transplant Int 1998; 11 (Suppl 1): 350-356

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant recipients in the Giessen renal transplant unit

Exclusion Criteria:

* Contraindications against blood-taking (anemia with hemoglobin<9.5 g/l, hypotension etc.)
* No informed consent by the patient

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 1998-01; Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Weimer, Prof. Dr., Principal Investigator — Department of Internal Medicine, University of Giessen, Germany
Locations (1):
- Department of Internal Medicine, University of Giessen, Giessen, Germany

REFERENCES:
- [Background] Weimer R, Mytilineos J, Feustel A, Preiss A, Daniel V, Grimm H, Wiesel M, Opelz G. Mycophenolate mofetil-based immunosuppression and cytokine genotypes: effects on monokine secretion and antigen presentation in long-term renal transplant recipients. Transplantation. 2003 Jun 27;75(12):2090-9. doi: 10.1097/01.TP.0000058808.37349.23. PMID 12829918
- [Background] Weimer R, Melk A, Daniel V, Friemann S, Padberg W, Opelz G. Switch from cyclosporine A to tacrolimus in renal transplant recipients: impact on Th1, Th2, and monokine responses. Hum Immunol. 2000 Sep;61(9):884-97. doi: 10.1016/s0198-8859(00)00152-x. PMID 11053632
- [Background] Weimer R, Zipperle S, Daniel V, Carl S, Staehler G, Opelz G. Superior 3-year kidney graft function in patients with impaired pretransplant Th2 responses. Transpl Int. 1998;11 Suppl 1:S350-6. doi: 10.1007/s001470050496. PMID 9665014
- [Background] Zipperle S, Weimer R, Golling M, Daniel V, Otto G, Opelz G. Impaired T-cell IL-10 secretion and CD4 helper function in liver transplant patients treated with tacrolimus. Transplant Proc. 1997 Feb-Mar;29(1-2):1079-80. doi: 10.1016/s0041-1345(96)00411-3. No abstract available. PMID 9123208
- [Background] Weimer R, Zipperle S, Daniel V, Carl S, Staehler G, Opelz G. Pretransplant CD4 helper function and interleukin 10 response predict risk of acute kidney graft rejection. Transplantation. 1996 Dec 15;62(11):1606-14. doi: 10.1097/00007890-199612150-00014. PMID 8970616
- [Background] Weimer R, Zipperle S, Daniel V, Pomer S, Staehler G, Opelz G. IL-6 independent monocyte/B cell defect in renal transplant recipients with long-term stable graft function. Transplantation. 1994 Jan;57(1):54-9. doi: 10.1097/00007890-199401000-00011. PMID 7507271
- [Result] Weimer R, Streller S, Staak A, Heilke M, Li D, Dietrich H, Daniel V, Feustel A, Rainer L, Zinn S, Friemann S, Ernst W, Grimm H, Padberg W, Zimmermann T, Opelz G. Effects of three immunosuppressive regimens on CD4 helper function, B cell monocyte and cytokine responses in renal transplant recipients: 4-month follow-up of a prospective randomized study. Transplant Proc. 2002 Sep;34(6):2377-8. doi: 10.1016/s0041-1345(02)03278-5. No abstract available. PMID 12270445
- [Result] Weimer R, Staak A, Susal C, Streller S, Yildiz S, Pelzl S, Renner F, Dietrich H, Daniel V, Rainer L, Kamali-Ernst S, Ernst W, Padberg W, Opelz G. ATG induction therapy: long-term effects on Th1 but not on Th2 responses. Transpl Int. 2005 Feb;18(2):226-36. doi: 10.1111/j.1432-2277.2004.00047.x. PMID 15691277
- [Result] Weimer R, Susal C, Yildiz S, Streller S, Pelzl S, Staak A, Renner F, Dietrich H, Daniel V, Feuring E, Kamali-Ernst S, Ernst W, Padberg W, Opelz G. sCD30 and neopterin as risk factors of chronic renal transplant rejection: impact of cyclosporine A, tacrolimus, and mycophenolate mofetil. Transplant Proc. 2005 May;37(4):1776-8. doi: 10.1016/j.transproceed.2005.02.088. PMID 15919463
- [Result] Weimer R, Susal C, Yildiz S, Staak A, Pelzl S, Renner F, Dietrich H, Daniel V, Kamali-Ernst S, Ernst W, Padberg W, Opelz G. Post-transplant sCD30 and neopterin as predictors of chronic allograft nephropathy: impact of different immunosuppressive regimens. Am J Transplant. 2006 Aug;6(8):1865-74. doi: 10.1111/j.1600-6143.2006.01407.x. Epub 2006 Jun 9. PMID 16771810
- [Derived] Weimer R, Ettrich M, Renner F, Dietrich H, Susal C, Deisz S, Padberg W, Opelz G. ATG induction in renal transplant recipients: Long-term hazard of severe infection is associated with long-term functional T cell impairment but not the ATG-induced CD4 cell decline. Hum Immunol. 2014 Jun;75(6):561-9. doi: 10.1016/j.humimm.2014.02.015. Epub 2014 Feb 12. PMID 24530759
- [Derived] Weimer R, Deisz S, Dietrich H, Renner F, Bodeker RH, Daniel V, Kamali-Ernst S, Ernst W, Padberg W, Opelz G. Impact of maintenance immunosuppressive regimens--balance between graft protective suppression of immune functions and a near physiological immune response. Transpl Int. 2011 Jun;24(6):596-609. doi: 10.1111/j.1432-2277.2011.01241.x. Epub 2011 Mar 14. PMID 21401729